CLINICAL TRIAL: NCT06592872
Title: Using Digital Health Technology to Prevent Bullying and Cyberbullying Among Elementary School Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Williams (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Christopher Williams, Senior Vice President, National Health Promotion Associates, Inc.
Organization: National Health Promotion Associates, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44HD114361 (NIH); R44HD114361 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Bullying; Cyberbullying; Smoking
Keywords: bullying; cyberbullying; elementary school; videogame; educational games
MeSH Terms: conditions — Bullying; Cyberbullying; Smoking

STUDY DESIGN:
Intervention Model Description: The intervention will consist of a suite of serious (educational) videogames and interactive teacher-led classroom sessions. The intervention is designed to address the urgent need for an effective primary prevention approach to the problem of bullying and cyberbullying among elementary school students. The intervention enhances personal self-management skills, social skills, refusal skills, and other life skills needed to successfully navigate developmental tasks, increase resilience, and facilitate healthy psychosocial development.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LifeSkills for Elementary School (Intervention) (Experimental): Approximately 1500 students in the 3rd grade (100 students per school) will complete pre-tests, post-tests, and 12- and 24-month follow-ups. Students whose school is randomized to the intervention condition (15 schools) will receive the LifeSkills Training standard curriculum plus bullying/cyberbullying classroom and serious game.
  Interventions: Behavioral: Bullying prevention
- LifeSkills for Elementary School (Control) (No Intervention): Approximately 1500 students in the 3rd grade (100 students per school) will complete pre-tests, post-tests, and 12- and 24-month follow-ups. Students whose school is randomized to the control condition (12 schools) will not receive the LifeSkills Training intervention, but will receive the health education content normally provided by their schools.

INTERVENTIONS:
Behavioral: Bullying prevention — The intervention utilizes a serious (educational) videogame and teacher-led, interactive class sessions. Students exposed to the intervention will learn to respond to in-person and online bullying from the perspectives of perpetrator, victim, and bystander. The intervention enhances personal self-management skills, social skills, refusal skills, and other life skills needed to successfully navigate developmental tasks, increase resilience, and facilitate healthy psychosocial development.
  Arms: LifeSkills for Elementary School (Intervention)

SUMMARY:
This project is designed to address the urgent need for an effective primary prevention approach to the problem of bullying and cyberbullying among elementary school students. The project involves developing, feasibility testing, and testing for the effectiveness an innovative new approach to the primary prevention of bullying utilizing both a serious (educational) videogame and facilitator-led, interactive class sessions. Using a cluster randomized controlled trial, the intervention will teach students how to respond to in-person and online bullying from the perspectives of perpetrator, victim, and bystander. The intervention enhances personal self-management skills, social skills, refusal skills, and other life skills needed to successfully navigate developmental tasks, increase resilience, and facilitate healthy psychosocial development. At the end of the initial intervention period, and at one- and two-year follow-ups, we will compare outcomes of students in the intervention and control groups with respect to changes in behaviors, norms, attitudes, and knowledge regarding bullying, cyberbullying, and substance use behavior.

DETAILED DESCRIPTION:
Bullying and cyberbullying are highly prevalent forms of aggressive behavior among youth of all ages and have a wide variety of negative social and mental health consequences. Bullying in all its forms involves persistent and intentional threatening, aggressive or verbally abusive behavior directed toward others at relative disadvantage. These behaviors share a similar set of risk and protective factors with early-stage substance use, therefore a single intervention approach may efficiently address both behaviors. Indeed, a fruitful way to extend the benefits of evidence-based prevention is to adapt the most effective interventions so they address shared and unique risk and protective factors for multiple related behaviors. The proposed SBIR Fast-Track application requests funding to develop and evaluate a multicomponent intervention to prevent bullying behavior by adapting the evidence-based Life Skills Training (LST) elementary school program. LST teaches youth personal self-management skills, social skills, drug refusal skills, and other life skills needed to successfully navigate key developmental tasks, increase resilience, and facilitate healthy psychosocial development. The LST program has been extensively tested and found to effectively prevent substance use in a series of randomized controlled trials with behavioral effects reported in over 30 peer-reviewed publications. The intervention for the proposed SBIR will teach young people how to respond to in-person and online bullying from the perspectives of perpetrator, victim, and bystander. We propose to develop: (1) bullying-specific classroom sessions to supplement the existing LST elementary school program; (2) an immersive serious (educational) video game to provide opportunities for students to apply life skills in preventing bullying and other high-risk situations in a gamified format; and, (3) e-learning modules that provide parents with strategies and resources to support anti-bullying lessons taught in school; and (4) e-learning modules for educators and support professionals that emphasize the importance of a school-wide anti-bullying approach that teaches prosocial behavior and encourages respect for peers. In Phase I, we will develop prototypes of bullying-specific classroom sessions, a video game level, and teacher and parent training materials to test them for feasibility, usability, and overall appeal. In Phase II, we will complete the development of all program materials and conduct a rigorous randomized controlled trial (RCT) of the prevention program. Elementary schools (N=30) will be randomized to either an intervention group that receives the prevention program or a treatment-as-usual control group that receives existing school health education. At the end of the initial intervention period, and at one- and two-year follow-ups, we will compare both groups with respect to changes in behaviors, norms, attitudes, and knowledge regarding bullying, cyberbullying, and substance use behavior.

Phase II Specific Aims

1. Develop the complete multicomponent primary prevention curriculum materials to prevent bullying and cyberbullying among elementary school students;
2. Conduct a rigorous RCT that randomizes 30 elementary schools into either an intervention or treatment-as-usual control condition to test the effectiveness of the intervention;
3. Analyze outcome data to assess the impact of the intervention on behaviors, norms, attitudes, and knowledge regarding bullying, cyberbullying, and substance use at the end of the initial intervention period, and at 12- and 24-month follow-up assessments;
4. Conduct a process evaluation to document and monitor all Phase II project activities;
5. Disseminate research findings to the scientific and practice communities;
6. Create a provider training mechanism to promote dissemination and sustainability of the intervention;
7. Based on our commercialization plan, implement a marketing strategy for the new primary prevention program aimed at elementary schools across the country.

ELIGIBILITY:
Inclusion Criteria: All students are eligible to participate in the intervention and complete the surveys.

Exclusion Criteria: All students are eligible to participate in the intervention and complete the surveys. Survey data will be excluded from the analysis for participants with significant cognitive impairment or severe learning disabilities, as designated by school personnel.

-

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Bullying/cyberbullying, norms, and attitudes at posttest | Posttest (within 2 weeks of completing final classroom session/videogame module)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding bullying and cyberbullying and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Bullying and cyberbullying, norms, and attitudes at 24-month followup | 24-month followup (within 24-25 months of completing the final classroom session and videogame module)
  The investigtors will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding bullying and cyberbullying and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and control group.
Bullying/cyberbullying, norms, and attitudes at baseline | Pretest (prior to participation in the first classroom session and videogame module of intervention)
  The investigators will asess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding bullying and cyberbullying and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Bullying and cyberbullying, norms, and attitudes at 12-month followup | 12-month followup (within 12-13 months of completing final classroom session and videogame module
  The investigators will assess key study variables including behaviors, norms, attitudes, and knowledge regarding bullying and cyberbullying and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.

SECONDARY OUTCOMES:
Bullying and cyberbullying, norms, and attitudes at pretest (prior to participating in the first classroom session and videogame module) | Pretest (prior to participation in the first classroom session and videogame module of intervention)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding substance use and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Bullying and cyberbullying, norms, and attitudes at posttest (within 2 weeks of completing final classroom session and videogame module) | Posttest (within 2 weeks of completing final classroom session and videogame module)
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding bullying and cyberbullying and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and control group.
Bullying and cyberbullying, norms, and attitudes at 12-month followup | 12-month followup (within 12-13 months of completing final classroom session and videogame module
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding substance use and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.
Bullying and cyberbullying, norms, and attitudes at 24-month followup | 24-month followup (within 24-25 months of completing final classroom session and videogame module
  The investigators will assess (via questionnaire) key study variables including behaviors, norms, attitudes, and knowledge regarding substance use and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Williams, PhD, MPH, Principal Investigator — National Health Promotion Associates

IPD SHARING:
Plan to Share IPD: No